CLINICAL TRIAL: NCT04774900
Title: The Influence of Standardization of Ambulance Equipment on the Speed of Medical Procedures Provision
Brief Title: Standardization of Ambulance Equipment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: David Peran (Other Government)
Responsible Party: Sponsor-Investigator, David Peran, Head of Education and Training Centre, Emergency Medical Service, Prague
Organization: Emergency Medical Service, Prague (Other Government)
Other Study IDs: ZZSHMP_002_2021
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Safety Issues
Keywords: quality and safety; emergency medical services; paramedics; equipment; standardisation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standardised: The procedures will be observed with standardized equipment placement.
  Interventions: Procedure: Administration of oxygen; Procedure: Administration of drug in a nebulizer; Procedure: Securing intravenous line; Procedure: Administration of IV drug; Procedure: Needle decompression of tension pneumothorax
- Modified: The procedures will be observed with modified equipment placement - placement according to older methodology or custom.
  Interventions: Procedure: Administration of oxygen; Procedure: Administration of drug in a nebulizer; Procedure: Securing intravenous line; Procedure: Administration of IV drug; Procedure: Needle decompression of tension pneumothorax

INTERVENTIONS:
Procedure: Administration of oxygen — Administration of high-flow oxygen via face mask to a high fidelity mannequin.
Procedure: Administration of drug in a nebulizer — Administration of bronchodilator via nebulizer mask to a high fidelity mannequin.
Procedure: Securing intravenous line — Securing an intravenous line at the forearm of high fidelity mannequin.
Procedure: Administration of IV drug — Administration of bronchodilator via IV line to a high fidelity mannequin.
Procedure: Needle decompression of tension pneumothorax — Needle decompression of tension pneumothorax on a high fidelity mannequin.

SUMMARY:
The aim of the research is to find out what effect the standardization of ambulance equipment has on the speed of performing specific medical procedures.

DETAILED DESCRIPTION:
The aim of the research is to find out what effect the standardization of ambulance equipment has on the speed of performing specific medical procedures. In two simulated scenarios, the times from the decision to execution of medical procedures will be measured. In the first scenario, the equipment is located in the standard way and the research participants know where it is located. In the second scenario, the equipment is placed elsewhere and participants do not have the opportunity to check the equipment before the scenario. For the statistical comparison the Student's T-test and Wilcoxon signed-rank test will be used. For analysis of variance will be used the ANOVA test and for more than two dependent selections the Friedman's ANOVA test will be used.

ELIGIBILITY:
Inclusion Criteria:

* consent to participate
* times of all procedures recorded
* all procedures provided in a correct way - in meaning of quality of the procedure

Exclusion Criteria:

* disagreement with participation
* not all procedures provided or not provided correctly

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Paramedics of the Prague Emergency Medical Services - bachelor or higher professional education as paramedics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Time | Through study completion, an average of 6 months and/or until 100 cases will be collected.
  Time from decision to execution

CONTACTS AND LOCATIONS:
Overall Officials: David Peran, Dr., Study Chair — Prague EMS; Miroslav Tejkl, MS, Study Director — Prague EMS; Roman Sýkora, Ph.D., Principal Investigator — EMS of Karlovy Vary Region; Metodej Renza, MD, Principal Investigator — 3rd Faculty of Medicine, Charles University in Prague; Jaroslav Pekara, Ph.D., Principal Investigator — Prague EMS
Locations (1):
- Prague Emergency Medical Services, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No